CLINICAL TRIAL: NCT05970679
Title: A Randomized, Double Blind, Parallel, Multi-center, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of DW1125 and DW1125A in Patient With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DW1125 and DW1125A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW1125-301
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hypercholesterolemia, Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DW1125 (Experimental): 1 Ezetimibe/Atorvastatin 10/5 mg tablet orally once daily
  Interventions: Drug: Ezetimibe/Atorvastatin 10/5 mg; Drug: DW1125A placebo; Drug: DW1125E placebo; Drug: DW1125A-1 placebo
- DW1125A (Experimental): 1 Atorvastatin 5 mg tablet orally once daily
  Interventions: Drug: Atorvastatin 5mg; Drug: DW1125 placebo; Drug: DW1125E placebo; Drug: DW1125A-1 placebo
- DW1125E (Placebo Comparator): 1 Ezetimibe 10mg tablet orally once daily
  Interventions: Drug: Ezetimibe 10mg; Drug: DW1125 placebo; Drug: DW1125A placebo; Drug: DW1125A-1 placebo
- DW1125A-1 (Placebo Comparator): 1 Atorvastatin 10mg tablet orally once daily
  Interventions: Drug: Atorvastatin 10mg; Drug: DW1125 placebo; Drug: DW1125A placebo; Drug: DW1125E placebo

INTERVENTIONS:
Drug: Ezetimibe/Atorvastatin 10/5 mg — DW1125
  Arms: DW1125
Drug: Atorvastatin 5mg — DW1125A
  Arms: DW1125A
Drug: Ezetimibe 10mg — DW1125E
  Other Names: Ezetrol Tab. 10mg
  Arms: DW1125E
Drug: Atorvastatin 10mg — DW1125A-1
  Other Names: Lipiwon Tab. 10mg
  Arms: DW1125A-1
Drug: DW1125 placebo — Ezetimibe/Atorvastatin 10/5 mg placebo
  Arms: DW1125A; DW1125A-1; DW1125E
Drug: DW1125A placebo — Atorvastatin 5mg placebo
  Arms: DW1125; DW1125A-1; DW1125E
Drug: DW1125E placebo — Ezetimibe 10mg placebo
  Arms: DW1125; DW1125A; DW1125A-1
Drug: DW1125A-1 placebo — Atorvastatin 10mg placebo
  Arms: DW1125; DW1125A; DW1125E

SUMMARY:
A Randomized, Double blind, Parallel, Multi-center, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of DW1125 and DW1125A in Patient with primary Hypercholesterolemia or Mixed Dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* Both gender, the person aged 19 or older
* Patients who are diagnosed with primary Hypercholesterolemia or Mixed Dyslipidemia
* LDL- C ≤ 250 mg/dL and TG < 500 mg/dL on fasting status

Exclusion Criteria:

* Patients with Myopathy, Rhabdomyolysis, Fibromyalgia, hereditary neuromuscular disorders or family history, or Creatine kinase(CK) ≥ 2 x Upper Limit of Normal(ULN) on Visit 1
* Patients with severe renal disorders, Estimated Flomerular Filtration Rate (eGFR) < 30 mL/min/1.73m^2 on Visit 1
* Patients with hepatic failure or active or chronic hepatobiliary diseases or aspartate transaminase (AST) or alanine aminotransferase (ALT) ≥ 2.0 x ULN on visit 1

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
% Change of LDL-C | 8 weeks
  % Change of LDL-C in week 8 from baseline

SECONDARY OUTCOMES:
% Change of LDL-C | 4 weeks
  % Change of LDL-C in week 4 from baseline
% Change of Lipid parameters | 4 weeks and 8 weeks
  % Change of Lipid parameters(TC, TG, HDL-C, Non-HDL-C, Apo A1, Apo B) in week 4 and week 8 respectively after administrating the treatment drugs
LDL-C goal achievement rates | 4 weeks and 8 weeks
  LDL-C goal achievement rates in week 4 and week 8 respectively after administrating the treatment drugs (goal achievement for LDL-C: low risk group: < 160 mg/dL, intermediate risk group: <130 mg/dL, high risk group: < 100 mg/dL, extreme risk group: < 70 mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea